CLINICAL TRIAL: NCT03696264
Title: Protein Requirements in Resistance-trained Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Daniel Moore, Assistant Professor, University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RTM
Record Dates: First submitted 2018-10-01; First posted 2018-10-04 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Healthy
Keywords: Protein Requirements

STUDY DESIGN:
Masking Description: Participants blinded to the protein dose consumed in a given metabolic trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Resistance-trained, adult males (Experimental): Subjects receive varying levels of amino acid intakes ranging from 0.2-3.0g/kg/d
  Interventions: Dietary Supplement: Amino acid intake

INTERVENTIONS:
Dietary Supplement: Amino acid intake — Amino acid intake will range between 0.2-3.0g/kg/d

SUMMARY:
In this study, the investigators will use the minimally invasive indicator amino acid oxidation (IAAO) technique to determine protein requirements in resistance-trained males. It is hypothesized that the present study will show that protein requirements for resistance-trained males are i) greater than the current recommended dietary allowance (RDA) for non-active individual's comparable estimates, and ii) greater than existing nitrogen balance-based estimates for resistance-training individuals.

DETAILED DESCRIPTION:
The adequate ingestion of dietary protein is the most critical nutritional factor to support the growth and maintenance of lean body mass across the lifespan. Currently, the World Health Organization/Food and Agricultural Organization (WHO/FAO) suggest that daily protein requirements in healthy, non-active adults are 0.8 g/kg/day. However, of primary interest in the present study is the impact that exercise has on the nutritional requirement for dietary protein in habitually active adults (e.g., individuals performing chronic resistance training). Protein requirements for individuals who participate in strength-based exercise training have been suggested to range from 1.2-1.7 g protein/kg/day (1), which equates to a 50-112% increase from the current RDA. The increased requirement in strength training populations may reflect the requirement for protein to repair and/or rebuild muscle tissue by promoting anabolism (2). Nutritional requirements for dietary protein in adults (both active and non-active) have traditionally been determined utilizing the antiquated and often erroneous nitrogen balance (NBAL) technique (3), which is prone to underestimating protein requirements and therefore provides challenges to making accurate nutritional recommendations (4). This observation that NBAL underestimates protein requirements in non-active individuals could suggest that protein requirements are much greater than the current World Health Organization recommendation of 0.8 g/kg/day, which was evaluated using the NBAL technique (3). As a result, there is a need to re-evaluate recommendations utilizing advanced stable isotope methodology in order to characterize how dietary protein needs may be modulated by physical activity. Recent studies using the minimally invasive indicator amino acid oxidation (IAAO) technique have suggested that protein requirements in young men are at least 50% higher than WHO/FAO guidelines based on NBAL data (4). Furthermore, resistance training has been reported to increase (according to NBAL methodology) protein requirements by up to 75% (6). Therefore, in this study, the investigators will use the IAAO technique to determine protein requirements in resistance-trained males. It is hypothesized that protein requirements for resistance-trained males will be i) greater than the current RDA for non-active individual's comparable estimates, and ii) greater than existing NBAL-based estimates for resistance-training individuals.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, male weight-trained individuals that have trained consistently for >1 year.
* 18-35 years old.
* Train each muscle group (i.e. chest, back, legs) at least twice a week.
* Body mass stable in last month
* Meets strength relative to body weight guidelines (see below)

Bench Press:

Males- body weight (kg)*1.25

Leg Press:

Males- body weight (kg)* 4.0

Exclusion Criteria:

* Inability to meet health and physical activity guidelines according to the Physical Activity Readiness Questionnaire
* Inability to adhere to any of the protocol guidelines (i.e. alcohol, caffeine consumption)
* Regular tobacco use
* Illicit drug use (e.g. growth hormone, testosterone, etc.) (screened by survey sheet for training log
* >1 month sedentary in the last 6 months prior to study participation
* >30 min of continuous cardio per exercise session
* BMI (Body Mass Index) > 35.
* Individual plans to increase or decrease body mass in the next 3 months
* Habitually ingests greater than or equal to 3g protein kg/bw/day
* Use of supplements such as creatine and beta-alanine in the last 30 days.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Phenylalanine excretion | Through study completion, an average of 1 year
  Expressed as µmol/kg/h; phenylalanine excretion is determined via breath enrichment of the oral tracer

SECONDARY OUTCOMES:
Phenylalanine rate of appearance | Through study completion, an average of 1 year
  In µmol/kg/h; phenylalanine rate of appearance is determined via urinary enrichment of the oral tracer
Net Protein Balance | Through study completion, an average of 1 year
  In µmol/kg/h; calculated as the difference between whole-body protein synthesis and protein breakdown

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R Moore, PhD, Principal Investigator — University of Toronto
Locations (1):
- Goldring Centre for High Performance Sport, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Thomas DT, Erdman KA, Burke LM. Position of the Academy of Nutrition and Dietetics, Dietitians of Canada, and the American College of Sports Medicine: Nutrition and Athletic Performance. J Acad Nutr Diet. 2016 Mar;116(3):501-528. doi: 10.1016/j.jand.2015.12.006. PMID 26920240
- [Background] Phillips SM. Protein requirements and supplementation in strength sports. Nutrition. 2004 Jul-Aug;20(7-8):689-95. doi: 10.1016/j.nut.2004.04.009. PMID 15212752
- [Background] Rand WM, Pellett PL, Young VR. Meta-analysis of nitrogen balance studies for estimating protein requirements in healthy adults. Am J Clin Nutr. 2003 Jan;77(1):109-27. doi: 10.1093/ajcn/77.1.109. PMID 12499330
- [Background] Humayun MA, Elango R, Ball RO, Pencharz PB. Reevaluation of the protein requirement in young men with the indicator amino acid oxidation technique. Am J Clin Nutr. 2007 Oct;86(4):995-1002. doi: 10.1093/ajcn/86.4.995. PMID 17921376
- [Background] Tarnopolsky MA, Atkinson SA, MacDougall JD, Chesley A, Phillips S, Schwarcz HP. Evaluation of protein requirements for trained strength athletes. J Appl Physiol (1985). 1992 Nov;73(5):1986-95. doi: 10.1152/jappl.1992.73.5.1986. PMID 1474076
- [Derived] Mazzulla M, Abou Sawan S, Williamson E, Hannaian SJ, Volterman KA, West DWD, Moore DR. Protein Intake to Maximize Whole-Body Anabolism during Postexercise Recovery in Resistance-Trained Men with High Habitual Intakes is Severalfold Greater than the Current Recommended Dietary Allowance. J Nutr. 2020 Mar 1;150(3):505-511. doi: 10.1093/jn/nxz249. PMID 31618421